CLINICAL TRIAL: NCT00813566
Title: Multi-Tracer PET Assessment of Primary Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI31335
Record Dates: First submitted 2008-12-16; First posted 2008-12-23 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Brain Tumors; Cancer
Keywords: cancer; imaging; PET scanning
MeSH Terms: conditions — Brain Neoplasms; Neoplasms | interventions — Fluorodeoxyglucose F18; alovudine; carbon-11 acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): All participants will receive multi-tracer PET scans at up to 3 time points: baseline, at the conclusion of standard of care chemoradiation, and at the time of documented recurrence within two years.
  Interventions: Drug: [18F]fluoro-2-deoxy-D-glucose (FDG); Drug: 3'-deoxy-3'-[18F]fluorothymidine (FLT); Drug: [15O]-H2O; Drug: [11C]Acetate

INTERVENTIONS:
Drug: [18F]fluoro-2-deoxy-D-glucose (FDG) — Brain scan with metabolic imaging tracer that aids in assessment, diagnosis, and staging of patients with cancer.
  Other Names: FDG; [18F]FDG; FDG-PET/CT
Drug: 3'-deoxy-3'-[18F]fluorothymidine (FLT) — Brain scan with a radiolabeled imaging agent for investigating cellular proliferation of tumors
  Other Names: [18F]FLT; FLT
Drug: [15O]-H2O — Brain scan with imaging agent to determine tumor blood flow
  Other Names: H2[15O]; [15O]water
Drug: [11C]Acetate — Brain scan with imaging agent to determine growth activity of tumor
  Other Names: [11C]ACE; ACE

SUMMARY:
The standard treatment approach for patients with high-grade primary brain tumors includes maximum feasible surgical resection, followed by 6 weeks of concurrent cranial irradiation and daily low-dose temozolomide chemotherapy, followed by 12 cycles of high-dose temozolomide administered for 5 consecutive days every 4 weeks [Stupp 2005]. Contrast-enhanced MRI is the current standard for evaluating the success of therapy and monitoring for tumor recurrence. MRI is typically obtained prior to initial surgery, within 24 hours after surgery, at the conclusions of cranial irradiation, and then every 8 weeks during temozolomide chemotherapy until evidence of recurrence. Despite this careful clinical and radiographic surveillance, and despite decades of research into the histologic and molecular classification of primary brain tumors, our ability to predict tumor behavior remains very limited. Some gliomas will result in overall survival times of only months, whereas other histologically-identical gliomas may yield survivals of years to decades [Carson 2007, Curran 1993, Lamborn 2004]. Current assessment of tumor response to therapy is also poor. Patients with complete radiographic response after cranial irradiation often progress rapidly post-irradiation. In contrast, some patients with enhancing masses at the end of chemoradiotherapy may respond dramatically to further chemotherapy alone, or the masses may even disappear in the absence of further therapy (so called "tumor pseudoprogression") [Chamberlain 2007]. This confounding situation demonstrates a need for better assessment of tumor response.

DETAILED DESCRIPTION:
Positron emission tomography (PET) is a molecular imaging modality that can probe various aspects of tumor function using a variety of radio-labeled imaging agents ("tracers"). Oncologic PET imaging has seen a dramatic rise in clinical utilization over the past decade for cancer detection, staging, and evaluating residual or recurrent disease following therapy. These clinical scans use the tracer [18F]fluoro-2-deoxy-D-glucose (FDG), which accumulates in cells in proportion to glucose (GLUT) transporter and hexokinase activity. FDG thus provides a measure of tissue glucose metabolism. Concurrent with this clinical growth, a number of other PET tracers have received significant attention in research for a variety of imaging targets. Of special interest are the tracers 3'-deoxy-3'-[18F]fluorothymidine (FLT), 1-[11C]-acetate (ACE), and [15O]water (H2O). The uptake, retention/washout, and ultimate biodistribution of these tracers are each related to different functional or molecular processes. As such, each can be used to probe a different aspect of tumor function: FLT directly assesses tumor proliferation, ACE provides a measure of tumor growth related to fatty acid and membrane synthesis, and H2O quantifies tumor perfusion.

OBJECTIVES:

This study has two primary objectives: a translational objective in which a new PET imaging technology will be translated from experimental development (with simulations and in animals) to the first use in human subjects; and an exploratory objective in which the complementary value of multiple PET tracers will be investigated. Each of these objective is described below, where the study design has been carefully setup to fulfill both objectives in the same study population.

The translational objective of this study is to implement and evaluate a new imaging technology for rapid, single-scan multi-tracer PET imaging of these tracers. Current PET technology prohibits imaging of more than one tracer in a single scan since the imaging signals from each tracer cannot be distinguished by normal techniques; as such, separate scans with each tracer currently need to be acquired hours or days apart. Our group has developed techniques and algorithms for recovering individual-tracer images from rapidly-acquired multi-tracer PET data using dynamic imaging techniques. These methods have been tested through extensive simulations and verified experimentally in a canine model with spontaneously-occurring tumors. Refinement of the methods with more advanced algorithms is ongoing. The patient imaging studies of this protocol will be implemented in two phases. In Phase A, separate single-tracer imaging of each tracer will be performed. The data from these scans will be co-registered and combined to "emulate" multi-tracer scans, which will then be processed by the multi-tracer signal-separation algorithms. This will permit a direct comparison of imaging biomarkers from multi-tracer vs. single-tracer scans for each tracer. Such comparison techniques have been established by the investigators and have been accepted by peer review for testing multi-tracer signal-separation algorithms. Once statistically-significant evidence is obtained that multi-tracer scans can accurately provide the same imaging biomarkers as separate single-tracer scans, the imaging will transition to Phase B-in which actual multi-tracer scans will be performed.

The objectives of this exploratory study is to preliminarily evaluate the complementary value of FDG, FLT, ACE, and H2O PET in patients with primary glial neoplasms. Multi-tracer PET profiles with these four tracers will be obtained in 20 patients with primary glial neoplasms at up to three timepoints: (1) at "baseline" prior to surgery or immediately after surgery providing a complete surgical resection was not possible and confirmed by a post-operative contrast MRI scan where residual tumor greater than 1.0 cm in diameter was present and prior to any tumor-directed therapy; (2) at the conclusions of the initial (~6-8 weeks) chemoradiotherapy; and (3) at the time of MRI-documented recurrence within 2 years. In addition, patients with a known primary brain tumor who have previously undergone treatment and have recurred based on standard clinical and imaging criteria will be eligible for the study. A number of quantitative and pseudo-quantitative imaging biomarkers for each tracer will be computed at each imaging timepoint, and the change in each biomarker between timepoints will also be computed. These data will be compared with clinical endpoints (survival, time to progression), and with tumor biologic information (histology, WHO grade, vascularity, Ki-67, vascular endothelial growth factor (VEGF), epidermal growth factor receptor (EGFR), p53) in cases when tumor tissue becomes available from standard care. These data will provide pilot information into the potential value of concurrent multiple PET biomarkers for predicting tumor behavior prior to the start of therapy, for improved prognostication, for more efficient and effective tumor surveillance, and/or for more appropriate assignment of patients to conventional, aggressive, or investigational therapies early in their clinical courses.

The driving hypothesis for the overall line of research is that multiple PET imaging biomarkers obtained in conjunction can provide improved image-guided personalized care of patients with primary glial neoplasms. The term "personalized care" is used here to broadly include the prediction of tumor behavior prior to the start of therapy, tumor surveillance, prognostication, and individualized assignment of patients to conventional, aggressive, or investigational therapies early in their clinical courses. This pilot project will obtain initial data on the value of these PET biomarkers for such image-guided personalized care.

Specific hypotheses to be tested include:

* HYPOTHESIS I a: Rapid, single-scan multi-tracer PET imaging can recover PET imaging biomarker information of each tracer that are not significantly different from those obtained from conventional, single-tracer scans of each tracer.
* HYPOTHESIS II b: Multi-tracer PET biomarkers, obtained in conjunction, are better able to predict tumor aggressiveness than individual-tracer biomarkers or conventional radiographic imaging.
* HYPOTHESIS III b: Multi-tracer PET biomarkers, obtained in conjunction, are better able to detect functional changes in tumor state that occur in response to therapy than individual-tracer biomarkers or conventional radiographic imaging.
* HYPOTHESIS IV b: Characterization of multiple aspects of tumor function (glucose metabolism, proliferation, membrane growth, and perfusion) provides new insight into tumor status that can guide selection of the most appropriate therapy.

a Sufficient statistical power is expected to be obtained under this protocol to validate the extensive simulations and experimental evaluations performed previously and concurrently with these patient imaging studies.

b Pilot data regarding these three hypotheses will be obtained in this work by studying the correlation of PET imaging biomarkers with clinical outcomes and tumor biologic information. Though high statistical power cannot be expected from the limited number of patients in this pilot study, underlying trends in the data will be identified, permitting the formulation of formal hypotheses to be tested in future rigorous trials.

ELIGIBILITY:
Inclusion Criteria:

Three different adult patient groups will be eligible for inclusion in this study:

* Group 1: Adult patients with compelling evidence of primary brain tumor based on clinical and MRI or CT imaging characteristics that have not yet received surgery, histological diagnosis, or any tumor-directed therapy. Such evidence will include: MRI or CT scan-documented mass lesion within the brain, accompanied by anatomically appropriate neurological signs and symptoms, in the absence of a probable competing diagnosis such as brain abscess or primary intracranial hematoma.
* Group 2: Newly diagnosed primary malignant brain tumors (WHO Grade II - IV glial-based tumors) who have not had a complete surgical resection and by contrast MRI or CT have residual tumor greater than 1.0 cm in diameter and will be receiving radiotherapy and/or chemotherapy.
* Group 3: Patients with probable or possible recurrent primary brain tumor as determined by standard clinical criteria or MRI or CT imaging. The abnormality must be greater than or equal to 1.0 cm in diameter by contrast MRI or CT or show changes on non-enhancing MRI sequences (T2 or FLAIR).

  * Patients must be 18 years or older for inclusion in this study. There is little experience with the safety of [18F]FLT in children, and the risks associated with radiation exposure may be increased for children under 18 years old as well.
  * Karnofsky performance status ≥ 60%.
  * Patients must document their willingness to be followed for at least 24 months after recruitment by signing informed consent documenting their agreement to have clinical endpoints and the results of histopathologic tissue analysis (when tissue becomes available from routine care) entered into a research database.
  * All patients, or their legal guardians, must sign a written informed consent and HIPAA authorization in accordance with institutional guidelines.
  * Determination of pregnancy status: Female patients that are not postmenopausal or surgically sterile will undergo a serum pregnancy test prior to each set of multi-tracer PET scans. A negative test will be necessary for such patients to undergo research PET imaging.
  * Pre-treatment laboratory tests for patients receiving [18F]FLT must be performed within 21 days prior to study entry. These must be less than 2.5 times below or above the upper or lower limit range for the respective laboratory test for entry into the study. In those instances where a baseline laboratory value is outside of this range, then such a patient will be ineligible for enrollment. For the follow-up scanning sessions after therapy has been instituted, laboratory testing will also be required due to the use of FLT. The patients have brain tumors and will receive various forms of therapy; therefore many routine laboratory tests may not be within the typical normal range. As such, a factor of 4.0 times above or below the upper or lower value for the normal range for any laboratory test will be used to determine the acceptable range for the 2nd and possible 3rd imaging timepoints. The baseline laboratory testing will include liver enzymes (ALT, aspartate aminotransferase (AST), alkaline phosphatase (ALK), LDH), bilirubin (total), serum electrolytes, complete blood count (CBC) with platelets and absolute neutrophil counts, prothrombin time, partial thromboplastin time, blood urea nitrogen (BUN), creatinine. Previous urinalysis abnormalities will not preclude the patient from being studied. For those patients receiving coumadin or another anticoagulant the upper limit for prothrombin time or partial thromboplastin time must not exceed 6 times the upper limit of the normal range.

Exclusion Criteria:

* Patients with clinically significant signs of uncal herniation, such as acute pupillary enlargement, rapidly developing motor changes (over hours), or rapidly decreasing level of consciousness, are not eligible.
* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals. Patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion.
* Patients who are pregnant or lactating or who suspect they might be pregnant. Serum pregnancy tests will be obtained prior to each set of multi-tracer PET scans in female patients that are not postmenopausal or surgically sterile.
* Adult patients who require monitored anesthesia for PET scanning.
* HIV positive patients due to the previous toxicity noted with FLT in this patient group.
* Patients who have undergone surgery or receive any previous tumor-directed therapy for their brain tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-11-12 (Actual); Primary Completion 2015-02-03 (Actual); Study Completion 2015-02-03 (Actual)

PRIMARY OUTCOMES:
Rapid, single-scan multi-tracer PET imaging can recover PET imaging biomarker information of each tracer that are not significantly different from those obtained from conventional, single-tracer scans of each tracer. | June 2014
Multi-tracer PET biomarkers, obtained in conjunction, are better able to predict tumor aggressiveness than individual-tracer biomarkers or conventional radiographic imaging. | June 2014
Multi-tracer PET biomarkers, obtained in conjunction, are better able to detect functional changes in tumor state that occur in response to therapy than individual-tracer biomarkers or conventional radiographic imaging. | June 2014
Characterization of multiple aspects of tumor function (glucose metabolism, proliferation, membrane growth, and perfusion) provides new insight into tumor status that can guide selection of the most appropriate therapy. | June 2014

CONTACTS AND LOCATIONS:
Overall Officials: John M Hoffman, MD, Principal Investigator — Huntsman Cancer Institute; Daniel Kadrmas, PhD, Study Chair — Huntsman Cancer Institute; Randy Jensen, MD,PhD, Study Chair — Huntsman Cancer Institute; Howard Colman, MD,PhD, Study Chair — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States